CLINICAL TRIAL: NCT02685241
Title: Monitoring of Biomarkers by Portable Breath Gas Sensors: an Exploratory Study
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Collaborators: Swiss Federal Institute of Technology (Other)
Responsible Party: Principal Investigator, Malcolm Kohler, Prof. Dr. med., University of Zurich
Other Study IDs: BASEC-Nr. PB-2016-00141
Record Dates: First submitted 2016-02-05; First posted 2016-02-18 (Estimated); Last update posted 2019-10-18 (Actual); Status verified 2019-10

CONDITIONS: General Population
Keywords: Exhaled breath; Biomarker

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- General population: General population

SUMMARY:
Breath analysis is a non-invasive procedure to detect and monitor diseases and it is particularly attractive for patients who have to routinely check biomarkers, such as diabetics (blood glucose) or end-stage renal disease patients (creatinine). Preliminary data in a small study with healthy subjects showed a high correlation between blood glucose levels and acetone. Therefore, the objective of this study is to correlate biomarkers (glucose level and creatinine, respectively) with the corresponding target breath components (acetone and NH3, respectively) detected by portable gas sensors in the general population and to assess possible predictive models for biomarker estimations from the corresponding target breath component and predictive models to estimate abnormal biomarker concentrations.

DETAILED DESCRIPTION:
Breath analysis is a non-invasive procedure to detect and monitor diseases and it is particularly attractive for patients who have to routinely check biomarkers, such as diabetics (blood glucose) or end-stage renal disease patients (creatinine). The proposed breath sensors analyse breath in real-time with on-line display of breath parameters, are portable, simple to operate, inexpensive and offer a sufficiently low limit of detection for the target breath markers, thus making them of high interest for daily clinical practice. Preliminary data in a small study with healthy subjects showed a high correlation between blood glucose levels and acetone.

The primary objective of this study is to correlate biomarkers (glucose level and creatinine, respectively) with the corresponding target breath components (acetone and NH3, respectively) detected by portable gas sensors in the general population. The secondary objectives of the study are to assess possible predictive models for biomarker estimations from the corresponding target breath component and predictive models to estimate abnormal biomarker concentrations.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Age ≥ 18 years

Exclusion Criteria:

* Moribund or severe disease prohibiting protocol adherence
* Physical or intellectual impairment precluding informed consent or protocol adherence
* Pregnant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: General population
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2019-10 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
The primary outcome will be the correlation between biomarkers (glucose levels and creatinine, respectively) and target breath components (acetone and NH3, respectively) detected by portable gas sensors | one hour, single measurement, no follow-up

SECONDARY OUTCOMES:
The assessment of possible predictive models for biomarker estimations (glucose levels and creatinine) from the corresponding target breath component (acetone and NH3) and predictive models to estimate the abnormal biomarker concentrations. | one hour, single measurement, no follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm Kohler, MD, Principal Investigator — University of Zurich
Locations (1):
- University Hospital Zurich, Division of Pneumology, Zurich, Canton of Zurich, Switzerland